CLINICAL TRIAL: NCT06952985
Title: Role of Gum Chewing in Post-operative Gut Motility After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Maryam Aslam (Other)
Collaborators: CMH Gujranwala (Unknown)
Responsible Party: Sponsor-Investigator, Dr Maryam Aslam, Head of Department Gynaecology and Obstetrics, Combined Military Hospital Gujranwala
Organization: Combined Military Hospital Gujranwala (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 275
Record Dates: First submitted 2025-04-20; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section; Gum Chewing; Gut Motility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A participants who were given chewing gum 6 hours after the surgery, three times a day (Active Comparator): In group A participants were given chewing gum 6 hours after the surgery, three times a day till passage of flatus
  Interventions: Dietary Supplement: Sugar free chew gum
- Group B participants who were kept nil per oral till bowel sounds were audible (Active Comparator): In group B, participants were managed as per standard routine protocol i.e. allowing oral when gut sound were audible
  Interventions: Other: Nil Per Oral

INTERVENTIONS:
Dietary Supplement: Sugar free chew gum — Chew gum has a role in ERAS protocol which is significant in early post operative recovery as compared to normal routine care methods
  Arms: Group A participants who were given chewing gum 6 hours after the surgery, three times a day
Other: Nil Per Oral — According to classic protocols patient were kept nil per oral till bowel sounds were audible
  Arms: Group B participants who were kept nil per oral till bowel sounds were audible

SUMMARY:
Many women deliver by caesarean section nowadays. The proportion of women who deliver by caesarean section ranges from 15% to over 50%, in some countries. After a caesarean section it is common for the bowel to stop working for several hours or days. Although this usually resolves by itself in a few days, it may be very uncomfortable. The retained gases and stools can cause the mother's belly to become swollen and painful with cramps and she may feel nauseated and vomit so she is not able to eat. She may need additional medications to ease these symptoms and her hospital discharge may be delayed. The use of medications that relieve pain during labour and painkillers following the surgery can also delay bowel function. Small intestine activity after abdominal operations returns to normal function within a few hours, gastric activity returns to normal within 24-48 hours, and colon activity returns to normal within 48-72 hours. Due to the delayed motility of the gastrointestinal system in the postoperative period, gas and secretions accumulate in the stomach and small and large intestines, which causes abdominal distension, nausea, vomiting, and pain, all of which negatively affect the comfort level of the patients. Chewing sugar-free gum after cesarean section can promote the early recovery of gastrointestinal function, but the side effects of chewing gum are still unclear, which needs more clinical, large sample and high-quality studies to further verify.

ELIGIBILITY:
Inclusion Criteria:

* Females of age 18-40 years
* Parity <5
* Presenting at gestational age ≥ 37 weeks,
* Undergoing cesarean section (as per operational definition) under spinal anesthesia

Exclusion Criteria:

* Females with history of chronic constipation (medical record)
* Females with obstructed labour, hypothyroidism (TSH>5IU)
* Females with intra operative complications such as bowel injury, history of gastrointestinal surgery, and water and electrolyte disturbances (on medical record), abnormal placenta (accrete, increta, previa, abruption)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females only
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Mean Time of Passage of First flatus | 06 Months
  In group A, females were given chewing gum 6 hours after the surgery, three times a day till passage of flatus. In group B, females were managed as per standard routine protocol i.e. allowing oral when bowel sounds are audible. Mean time of passage of first flatus since procedure was noted in terms of hours.

SECONDARY OUTCOMES:
Mean Duration of Hospital Stay | 06 Months
  In both groups mean duration of hospital stay was noted in terms number of days required to stay in the hospital after cesarean. Patients were discharged once they were pain free and on oral medication.

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No